CLINICAL TRIAL: NCT00483249
Title: Endovascular Exclusion of Thoracoabdominal And/or Paravisceral Abdominal Aortic Aneurysm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Warren J. Gasper, MD (Other)
Responsible Party: Sponsor-Investigator, Warren J. Gasper, MD, Associate Professor, Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02810
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Paravisceral Abdominal Aortic Aneurysm
Keywords: Thoracoabdominal; Paravisceral; Aneurysm; Endovascular; Stent-Graft; Aorta
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): Endovascular Branched Stent-Graft: The investigational operation is done making small incisions in both groins and the right arm and placing a graft in the aorta through tubes that are inserted through the femoral and brachial arteries, than fastening it in position with metal springs(stents).
  Interventions: Device: Endovascular Branched Stent-Graft

INTERVENTIONS:
Device: Endovascular Branched Stent-Graft — Industry manufactured branched stent-graft for treatment of TAAA/PVAAA.

SUMMARY:
This is a study to assess the safety and effectiveness of endovascular treatment of thoracoabdominal (TAAA) and paravisceral abdominal (PVAAA) aortic aneurysms. The investigational operation involves placing a stent-graft over the aortic aneurysm.

DETAILED DESCRIPTION:
A TAAA or PVAAA is an abnormal enlargement of the aorta, the main artery in the chest and abdomen. The standard operation for TAAA of PVAAA is performed through a long incision extending down the side of the chest and the front of the abdomen. In the standard operation, the weak area of the aorta is replaced with a fabric sleeve (graft). The investigational operation is done making small incisions in both groins and the right arm and placing a graft in the aorta through tubes that are inserted through the femoral and brachial arteries, than fastening it in position with metal springs(stents). The combination of a stent and a graft is known as a stent-graft. Compared with standard operation, the potential advantages of endovascular TAAA/PVAAA repair include less pain, less disturbance of intestinal function, a lower risk of pulmonary or cardiac complications and shorter hospital stay. The main disadvantage of endovascular TAAA/PVAAA is an unknown success rate.

ELIGIBILITY:
Inclusion Criteria

1. Aortic aneurysms:

   * greater than or equal to 6 cm in diameter in men,
   * greater than or equal to 5.5 cm in diameter in women,
   * and/or larger than 5 cm in diameter and enlarging at a rate of more than 5 mm/year,
   * and/or iliac aneurysms larger than 4 cm in diameter.
2. Anticipated mortality comparable to published rates with conventional surgical treatment.
3. Life expectancy more than 2 years.
4. Ability to give informed consent.
5. Willingness to comply with follow-up schedule.
6. Suitable arterial anatomy for endovascular repair.

Exclusion Criteria

1. Free rupture of the aneurysm.
2. Pregnancy.
3. Known allergy to Nitinol, stainless steel, or polyester.
4. Unwillingness or inability to comply with the follow up schedule.
5. Serious systemic or groin infection.
6. Uncorrectable coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-05; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful implantation of TAAA branched stent-graft. | 1 month

SECONDARY OUTCOMES:
Long term success of TAAA branched stent-graft treatment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Warren J Gasper, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Division of Vascular Surgery, SFVAMC, San Francisco, California
  - Division of Vascular Surgery, UCSF, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford ES, DeNatale RW. Thoracoabdominal aortic aneurysm: observations regarding the natural course of the disease. J Vasc Surg. 1986 Apr;3(4):578-82. doi: 10.1067/mva.1986.avs0030578. PMID 3959256
- [Background] Svensson LG, Crawford ES, Hess KR, Coselli JS, Safi HJ. Experience with 1509 patients undergoing thoracoabdominal aortic operations. J Vasc Surg. 1993 Feb;17(2):357-68; discussion 368-70. PMID 8433431
- [Background] Martin GH, O'Hara PJ, Hertzer NR, Mascha EJ, Krajewski LP, Beven EG, Clair DG, Ouriel K. Surgical repair of aneurysms involving the suprarenal, visceral, and lower thoracic aortic segments: early results and late outcome. J Vasc Surg. 2000 May;31(5):851-62. doi: 10.1067/mva.2000.106481. PMID 10805874
- [Background] Cambria RP, Davison JK, Carter C, Brewster DC, Chang Y, Clark KA, Atamian S. Epidural cooling for spinal cord protection during thoracoabdominal aneurysm repair: A five-year experience. J Vasc Surg. 2000 Jun;31(6):1093-102. doi: 10.1067/mva.2000.106492. PMID 10842145
- [Background] Walker SR, Yusuf SW, Wenham PW, Hopkinson BR. Renal complications following endovascular repair of abdominal aortic aneurysms. J Endovasc Surg. 1998 Nov;5(4):318-22. doi: 10.1583/1074-6218(1998)0052.0.CO;2. PMID 9867320
- [Background] Thompson JP, Boyle JR, Thompson MM, Strupish J, Bell PR, Smith G. Cardiovascular and catecholamine responses during endovascular and conventional abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 1999 Apr;17(4):326-33. doi: 10.1053/ejvs.1998.0760. PMID 10204055
- [Background] Zarins CK, White RA, Schwarten D, Kinney E, Diethrich EB, Hodgson KJ, Fogarty TJ. AneuRx stent graft versus open surgical repair of abdominal aortic aneurysms: multicenter prospective clinical trial. J Vasc Surg. 1999 Feb;29(2):292-305; discussion 306-8. doi: 10.1016/s0741-5214(99)70382-4. PMID 9950987
- [Background] May J, White GH, Yu W, Ly CN, Waugh R, Stephen MS, Arulchelvam M, Harris JP. Concurrent comparison of endoluminal versus open repair in the treatment of abdominal aortic aneurysms: analysis of 303 patients by life table method. J Vasc Surg. 1998 Feb;27(2):213-20; discussion 220-1. doi: 10.1016/s0741-5214(98)70352-0. PMID 9510276
- [Background] Chuter TA, Reilly LM, Faruqi RM, Kerlan RB, Sawhney R, Canto CJ, LaBerge JM, Wilson MW, Gordon RL, Wall SD, Rapp J, Messina LM. Endovascular aneurysm repair in high-risk patients. J Vasc Surg. 2000 Jan;31(1 Pt 1):122-33. doi: 10.1016/s0741-5214(00)70074-7. PMID 10642715
- [Background] Mitchell RS, Miller DC, Dake MD, Semba CP, Moore KA, Sakai T. Thoracic aortic aneurysm repair with an endovascular stent graft: the "first generation". Ann Thorac Surg. 1999 Jun;67(6):1971-4; discussion 1979-80. doi: 10.1016/s0003-4975(99)00436-1. PMID 10391350
- [Background] Kinney EV, Kaebnick HW, Mitchell RA, Jung MT. Repair of mycotic paravisceral aneurysm with a fenestrated stent-graft. J Endovasc Ther. 2000 Jun;7(3):192-7. doi: 10.1177/152660280000700304. PMID 10883955
- [Background] Iwase T, Inoue K, Sato M, Yoshida Y, Ueno K, Tanaka H, Tamaki S. Transluminal repair of an infrarenal aortoiliac aneurysm by a combination of bifurcated and branched stent grafts. Catheter Cardiovasc Interv. 1999 Aug;47(4):491-4. doi: 10.1002/(SICI)1522-726X(199908)47:43.0.CO;2-I. PMID 10470482
- [Background] Chuter TA, Gordon RL, Reilly LM, Goodman JD, Messina LM. An endovascular system for thoracoabdominal aortic aneurysm repair. J Endovasc Ther. 2001 Feb;8(1):25-33. doi: 10.1177/152660280100800104. PMID 11220464
- [Background] Anderson JL, Berce M, Hartley DE. Endoluminal aortic grafting with renal and superior mesenteric artery incorporation by graft fenestration. J Endovasc Ther. 2001 Feb;8(1):3-15. doi: 10.1177/152660280100800102. PMID 11220465
- [Background] Chuter TA, Buck DG, Schneider DB, Reilly LM, Messina LM. Development of a branched stent-graft for endovascular repair of aortic arch aneurysms. J Endovasc Ther. 2003 Oct;10(5):940-5. doi: 10.1177/152660280301000517. PMID 14656176
- [Background] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Background] Chuter TA, Hiramoto JS, Park KH, Reilly LM. The transition from custom-made to standardized multibranched thoracoabdominal aortic stent grafts. J Vasc Surg. 2011 Sep;54(3):660-7; discussion 667-8. doi: 10.1016/j.jvs.2011.03.005. Epub 2011 Jul 23. PMID 21788114
- [Background] Chuter T, Greenberg RK. Standardized off-the-shelf components for multibranched endovascular repair of thoracoabdominal aortic aneurysms. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):195-201. doi: 10.1177/1531003511430397. PMID 22205654
- [Background] Reilly LM, Rapp JH, Grenon SM, Hiramoto JS, Sobel J, Chuter TA. Efficacy and durability of endovascular thoracoabdominal aortic aneurysm repair using the caudally directed cuff technique. J Vasc Surg. 2012 Jul;56(1):53-63; discussion 63-4. doi: 10.1016/j.jvs.2012.01.006. Epub 2012 May 3. PMID 22560233
- [Background] Gasper WJ, Reilly LM, Rapp JH, Grenon SM, Hiramoto JS, Sobel JD, Chuter TA. Assessing the anatomic applicability of the multibranched endovascular repair of thoracoabdominal aortic aneurysm technique. J Vasc Surg. 2013 Jun;57(6):1553-8; discussion 1558. doi: 10.1016/j.jvs.2012.12.021. Epub 2013 Feb 6. PMID 23395201
- [Background] Premprabha D, Sobel J, Pua C, Chong K, Reilly LM, Chuter TA, Hiramoto JS. Visceral branch occlusion following aneurysm repair using multibranched thoracoabdominal stent-grafts. J Endovasc Ther. 2014 Dec;21(6):783-90. doi: 10.1583/14-4807R.1. PMID 25453879
- [Background] Sobel JD, Vartanian SM, Gasper WJ, Hiramoto JS, Chuter TA, Reilly LM. Lower extremity weakness after endovascular aneurysm repair with multibranched thoracoabdominal stent grafts. J Vasc Surg. 2015 Mar;61(3):623-8. doi: 10.1016/j.jvs.2014.10.013. Epub 2014 Nov 25. PMID 25457458
- [Background] Fernandez CC, Sobel JD, Gasper WJ, Vartanian SM, Reilly LM, Chuter TA, Hiramoto JS. Standard off-the-shelf versus custom-made multibranched thoracoabdominal aortic stent grafts. J Vasc Surg. 2016 May;63(5):1208-15. doi: 10.1016/j.jvs.2015.11.035. Epub 2016 Jan 24. PMID 26817612
- [Background] Ramanan B, Fernandez CC, Sobel JD, Gasper WJ, Vartanian SM, Reilly LM, Chuter TA, Hiramoto JS. Low-profile versus standard-profile multibranched thoracoabdominal aortic stent grafts. J Vasc Surg. 2016 Jul;64(1):39-45. doi: 10.1016/j.jvs.2016.01.038. Epub 2016 Mar 22. PMID 26994953
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Derived] Werlin EC, Kaushik S, Gasper WJ, Hoffman M, Reilly LM, Chuter TA, Hiramoto JS. Multibranched endovascular aortic aneurysm repair in patients with and without chronic aortic dissections. J Vasc Surg. 2019 Nov;70(5):1419-1426. doi: 10.1016/j.jvs.2019.02.048. Epub 2019 Jul 18. PMID 31327618
- [Derived] Walker J, Kaushik S, Hoffman M, Gasper W, Hiramoto J, Reilly L, Chuter T. Long-term durability of multibranched endovascular repair of thoracoabdominal and pararenal aortic aneurysms. J Vasc Surg. 2019 Feb;69(2):341-347. doi: 10.1016/j.jvs.2018.04.074. PMID 30683193
- [Derived] Chang CK, Chuter TA, Niemann CU, Shlipak MG, Cohen MJ, Reilly LM, Hiramoto JS. Systemic inflammation, coagulopathy, and acute renal insufficiency following endovascular thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2009 May;49(5):1140-6. doi: 10.1016/j.jvs.2008.11.102. PMID 19394543